CLINICAL TRIAL: NCT04539704
Title: Assessing Impacts of Static Magnetic Fields on Peripheral Pulses and Skin Blood Flow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Responsible Party: Principal Investigator, Harvey N. Mayrovitz, PhD, Professor, Nova Southeastern University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 2019-598-NSU
Record Dates: First submitted 2020-08-31; First posted 2020-09-07 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Arterial Stiffness; Magnetic Field Exposure; Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Subjects and coinvestigators making measurements are blinded to which devices are the active magnets and which are the sham magnets. Only the PI will have that information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Healthy Adults-magnet (Experimental): Healthy adults with magnet and/or sham
  Interventions: Device: magnet and sham
- Healthy Adults-sham (Sham Comparator): Healthy adults with magnet and/or sham
  Interventions: Device: magnet and sham

INTERVENTIONS:
Device: magnet and sham — In same subject some areas will have magnet and others will have sham

SUMMARY:
The purpose of this research study is to investigate and determine the effects of static magnetic fields produced by a small magnet on peripheral pulses and skin blood flow.

DETAILED DESCRIPTION:
A specific neodymium magnet and sham device will be placed on certain sites near the ulnar and medial arteries and the effect of such placement on peripheral pulses assessed via PPG on fingers and on skin blood flow via laser Doppler perfusion determined. These assessments will be made while healthy subjects are lying supine on a padded examination table over a time interval of about 45-60 minutes. In addition to the impact that either the magnet or the sham devices have, the pulse and skin blood flow patterns and features will be analyzed from the point of view of sequential variability with and eye toward developing related parameters to potentially improve such variability.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-35 years
2. No known neurological deficit
3. No known cardiovascular condition

Exclusion Criteria:

1. Unable or unwilling to lie reasonably still for about 55 minutes
2. Known to have diabetes of any type
3. Having any metallic or wire implant

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Effect of magnet on skin blood flow | one hour
  skin blood flow
Effect of magnet on arterial pulses | one hour
  Pulse values and paterns
Characterization of temporal pattern of pulse changes and their amelioration | one hour
  variability with and without normalization

CONTACTS AND LOCATIONS:
Locations (1):
- Nova Southeastern University, Davie, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mayrovitz HN, Astudillo A, Shams E. Finger skin blood perfusion during exposure of ulnar and median nerves to the static magnetic field of a rare-earth magnet: A randomized pilot study. Electromagn Biol Med. 2021 Jan 2;40(1):1-10. doi: 10.1080/15368378.2020.1856682. Epub 2020 Dec 5. PMID 33283550